CLINICAL TRIAL: NCT05555550
Title: Evaluation of 18F-Fluciclovine PET-MRI as a Biomarker of Response in Pediatric and Young Adult Patients With Low Grade Gliomas (LGG)
Brief Title: Evaluation of 18F-Fluciclovine Positron Emission Tomography - Magnetic Resonance Imaging (PET-MRI) in LGG
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Blue Earth Diagnostics (Industry); Dragon Master Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-019390; 21NO104 (Other: CHOP)
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Glioma; Low-grade Glioma; Low Grade Glioma of Brain; Glioma, Malignant; Glioma Intracranial
Keywords: Glioma; Low-grade Glioma; Low Grade Glioma of Brain; Glioma, Malignant; Glioma Intracranial; 18F-Fluciclovine
MeSH Terms: conditions — Glioma | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-Fluciclovine (Experimental): 18F-Fluciclovine PET-MRI
  Interventions: Drug: 18F-Fluciclovine

INTERVENTIONS:
Drug: 18F-Fluciclovine — 18F-Fluciclovine will be injected via IV prior to PET-MRI imaging
  Other Names: Axumin

SUMMARY:
The purpose of this study is to see if 18F-Fluciclovine (Axumin®) is useful and safe in the management of children with Low Grade Gliomas (LGG). Imaging with 18F-Fluciclovine PET-MRI will be performed prior to initiation of therapy for LGG, and then 3 months, and 1 year after starting therapy. Changes in 18F-Fluciclovine uptake will be compared to changes in MRI measurements at 3 months and 1 year as compared to baseline.

ELIGIBILITY:
Inclusion Criteria

1. LGG including the brainstem and supratentorial only (WHO grade I-II), confirmed by biopsy unless in NF1 participants with classic appearance.
2. Participants must have evaluable disease (1x1 cm tumor on MRI)
3. Scheduled to receive systemic therapy for LGG
4. Performance Score: Karnofsky ≥ 50 for participants > 16 years of age and Lansky ≥ 50 for participants ≤ 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Age: Participants must be ≥ 1 years but ≤21 years of age at registration
6. Being on a treatment regimen does not exclude a subject from enrollment.

Exclusion Criteria

1. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
2. Pregnant participants
3. Participants who weigh less than 8 kg.
4. Participants who cannot avoid contact with a pregnant woman or infant for at least 12 hours following injection.
5. Participants with a history of abnormal kidney function or creatinine >= CTCAE v5.0 grade 2 at time of study registration.
6. Participants with primary tumors of the spinal cord.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Compare change in standardized uptake value parameters (SUVmax and SUVpeak) on metabolic tumor volume in 18F-Fluciclovine PET | 1 year
  To identify change in the standardized uptake value (SUV) parameters (SUVmax, SUVpeak) for the 18F-Fluciclovine PET scan
Compare changes in pretreatment tumor measurement on MRI in pediatric participants who initiate systemic treatment for LGG | 1 year
  Calculate the change in tumor measurement on MRI

SECONDARY OUTCOMES:
Safety of 18F-Fluciclovine | 13 months
  The Safety profile of 18F-Fluciclovine PET in pediatric LGG participants will be accessed by the CTCAE 5.0 toxicity experienced after administration of 18F-Fluciclovine

OTHER OUTCOMES:
Response prediction | 1 year
  Determine if Baseline PET uptake as predictors of treatment response
Disease Progression | 1 year
  Identify changes in PET metrics at the time of progression

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Aboian, MD,PhD, Principal Investigator — The Children s Hospital of Philadelphia
Locations (1):
- The Children s Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones DTW, Kieran MW, Bouffet E, Alexandrescu S, Bandopadhayay P, Bornhorst M, Ellison D, Fangusaro J, Fisher MJ, Foreman N, Fouladi M, Hargrave D, Hawkins C, Jabado N, Massimino M, Mueller S, Perilongo G, Schouten van Meeteren AYN, Tabori U, Warren K, Waanders AJ, Walker D, Weiss W, Witt O, Wright K, Zhu Y, Bowers DC, Pfister SM, Packer RJ. Pediatric low-grade gliomas: next biologically driven steps. Neuro Oncol. 2018 Jan 22;20(2):160-173. doi: 10.1093/neuonc/nox141. PMID 29016845
- [Background] de Blank P, Bandopadhayay P, Haas-Kogan D, Fouladi M, Fangusaro J. Management of pediatric low-grade glioma. Curr Opin Pediatr. 2019 Feb;31(1):21-27. doi: 10.1097/MOP.0000000000000717. PMID 30531227
- [Background] Fangusaro J, Onar-Thomas A, Young Poussaint T, Wu S, Ligon AH, Lindeman N, Banerjee A, Packer RJ, Kilburn LB, Goldman S, Pollack IF, Qaddoumi I, Jakacki RI, Fisher PG, Dhall G, Baxter P, Kreissman SG, Stewart CF, Jones DTW, Pfister SM, Vezina G, Stern JS, Panigrahy A, Patay Z, Tamrazi B, Jones JY, Haque SS, Enterline DS, Cha S, Fisher MJ, Doyle LA, Smith M, Dunkel IJ, Fouladi M. Selumetinib in paediatric patients with BRAF-aberrant or neurofibromatosis type 1-associated recurrent, refractory, or progressive low-grade glioma: a multicentre, phase 2 trial. Lancet Oncol. 2019 Jul;20(7):1011-1022. doi: 10.1016/S1470-2045(19)30277-3. Epub 2019 May 28. PMID 31151904
- [Background] Ater JL, Xia C, Mazewski CM, Booth TN, Freyer DR, Packer RJ, Sposto R, Vezina G, Pollack IF. Nonrandomized comparison of neurofibromatosis type 1 and non-neurofibromatosis type 1 children who received carboplatin and vincristine for progressive low-grade glioma: A report from the Children's Oncology Group. Cancer. 2016 Jun 15;122(12):1928-36. doi: 10.1002/cncr.29987. Epub 2016 Apr 8. PMID 27061921
- [Background] Songmen S, Nepal P, Olsavsky T, Sapire J. Axumin Positron Emission Tomography: Novel Agent for Prostate Cancer Biochemical Recurrence. J Clin Imaging Sci. 2019 Nov 6;9:49. doi: 10.25259/JCIS_139_2019. eCollection 2019. PMID 31819826
- [Background] Wakabayashi T, Iuchi T, Tsuyuguchi N, Nishikawa R, Arakawa Y, Sasayama T, Miyake K, Nariai T, Narita Y, Hashimoto N, Okuda O, Matsuda H, Kubota K, Ito K, Nakazato Y, Kubomura K. Diagnostic Performance and Safety of Positron Emission Tomography Using 18F-Fluciclovine in Patients with Clinically Suspected High- or Low-grade Gliomas: A Multicenter Phase IIb Trial. Asia Ocean J Nucl Med Biol. 2017 Winter;5(1):10-21. doi: 10.22038/aojnmb.2016.7869. PMID 28840134
- [Background] Shoup TM, Olson J, Hoffman JM, Votaw J, Eshima D, Eshima L, Camp VM, Stabin M, Votaw D, Goodman MM. Synthesis and evaluation of [18F]1-amino-3-fluorocyclobutane-1-carboxylic acid to image brain tumors. J Nucl Med. 1999 Feb;40(2):331-8. PMID 10025843
- [Background] Michaud L, Beattie BJ, Akhurst T, Dunphy M, Zanzonico P, Finn R, Mauguen A, Schoder H, Weber WA, Lassman AB, Blasberg R. 18F-Fluciclovine (18F-FACBC) PET imaging of recurrent brain tumors. Eur J Nucl Med Mol Imaging. 2020 Jun;47(6):1353-1367. doi: 10.1007/s00259-019-04433-1. Epub 2019 Aug 15. PMID 31418054
- [Background] Tsuyuguchi N, Terakawa Y, Uda T, Nakajo K, Kanemura Y. Diagnosis of Brain Tumors Using Amino Acid Transport PET Imaging with 18F-fluciclovine: A Comparative Study with L-methyl-11C-methionine PET Imaging. Asia Ocean J Nucl Med Biol. 2017 Spring;5(2):85-94. doi: 10.22038/aojnmb.2017.8843. PMID 28660218
- [Background] Parent EE, Benayoun M, Ibeanu I, Olson JJ, Hadjipanayis CG, Brat DJ, Adhikarla V, Nye J, Schuster DM, Goodman MM. [18F]Fluciclovine PET discrimination between high- and low-grade gliomas. EJNMMI Res. 2018 Jul 25;8(1):67. doi: 10.1186/s13550-018-0415-3. PMID 30046944
- [Background] Kondo A, Ishii H, Aoki S, Suzuki M, Nagasawa H, Kubota K, Minamimoto R, Arakawa A, Tominaga M, Arai H. Phase IIa clinical study of [18F]fluciclovine: efficacy and safety of a new PET tracer for brain tumors. Ann Nucl Med. 2016 Nov;30(9):608-618. doi: 10.1007/s12149-016-1102-y. Epub 2016 Jul 14. PMID 27418267
- [Background] Liu CJ, Lu MY, Liu YL, Ko CL, Ko KY, Tzen KY, Chang HH, Yang YL, Jou ST, Hsu WM, Yen RF. Risk Stratification of Pediatric Patients With Neuroblastoma Using Volumetric Parameters of 18F-FDG and 18F-DOPA PET/CT. Clin Nucl Med. 2017 Mar;42(3):e142-e148. doi: 10.1097/RLU.0000000000001529. PMID 28072621
- [Background] Marner L, Nysom K, Sehested A, Borgwardt L, Mathiasen R, Henriksen OM, Lundemann M, Munck Af Rosenschold P, Thomsen C, Bogeskov L, Skjoth-Rasmussen J, Juhler M, Kruse A, Broholm H, Scheie D, Lauritsen T, Forman JL, Wehner PS, Hojgaard L, Law I. Early Postoperative 18F-FET PET/MRI for Pediatric Brain and Spinal Cord Tumors. J Nucl Med. 2019 Aug;60(8):1053-1058. doi: 10.2967/jnumed.118.220293. Epub 2019 Jan 25. PMID 30683767
- [Background] Morana G, Piccardo A, Puntoni M, Nozza P, Cama A, Raso A, Mascelli S, Massollo M, Milanaccio C, Garre ML, Rossi A. Diagnostic and prognostic value of 18F-DOPA PET and 1H-MR spectroscopy in pediatric supratentorial infiltrative gliomas: a comparative study. Neuro Oncol. 2015 Dec;17(12):1637-47. doi: 10.1093/neuonc/nov099. Epub 2015 Sep 23. PMID 26405202
- [Background] Albert NL, Weller M, Suchorska B, Galldiks N, Soffietti R, Kim MM, la Fougere C, Pope W, Law I, Arbizu J, Chamberlain MC, Vogelbaum M, Ellingson BM, Tonn JC. Response Assessment in Neuro-Oncology working group and European Association for Neuro-Oncology recommendations for the clinical use of PET imaging in gliomas. Neuro Oncol. 2016 Sep;18(9):1199-208. doi: 10.1093/neuonc/now058. Epub 2016 Apr 21. PMID 27106405
- [Background] Werner JM, Lohmann P, Fink GR, Langen KJ, Galldiks N. Current Landscape and Emerging Fields of PET Imaging in Patients with Brain Tumors. Molecules. 2020 Mar 24;25(6):1471. doi: 10.3390/molecules25061471. PMID 32213992
- [Background] Bhutia YD, Babu E, Ramachandran S, Ganapathy V. Amino Acid transporters in cancer and their relevance to "glutamine addiction": novel targets for the design of a new class of anticancer drugs. Cancer Res. 2015 May 1;75(9):1782-8. doi: 10.1158/0008-5472.CAN-14-3745. Epub 2015 Apr 8. PMID 25855379
- [Background] Galldiks N, Law I, Pope WB, Arbizu J, Langen KJ. The use of amino acid PET and conventional MRI for monitoring of brain tumor therapy. Neuroimage Clin. 2016 Dec 18;13:386-394. doi: 10.1016/j.nicl.2016.12.020. eCollection 2017. PMID 28116231
- [Background] Morana G, Piccardo A, Tortora D, Puntoni M, Severino M, Nozza P, Ravegnani M, Consales A, Mascelli S, Raso A, Cabria M, Verrico A, Milanaccio C, Rossi A. Grading and outcome prediction of pediatric diffuse astrocytic tumors with diffusion and arterial spin labeling perfusion MRI in comparison with 18F-DOPA PET. Eur J Nucl Med Mol Imaging. 2017 Nov;44(12):2084-2093. doi: 10.1007/s00259-017-3777-2. Epub 2017 Jul 27. PMID 28752225
- [Background] Dunkl V, Cleff C, Stoffels G, Judov N, Sarikaya-Seiwert S, Law I, Bogeskov L, Nysom K, Andersen SB, Steiger HJ, Fink GR, Reifenberger G, Shah NJ, Coenen HH, Langen KJ, Galldiks N. The usefulness of dynamic O-(2-18F-fluoroethyl)-L-tyrosine PET in the clinical evaluation of brain tumors in children and adolescents. J Nucl Med. 2015 Jan;56(1):88-92. doi: 10.2967/jnumed.114.148734. Epub 2014 Dec 18. PMID 25525183
- [Background] Galldiks N, Niyazi M, Grosu AL, Kocher M, Langen KJ, Law I, Minniti G, Kim MM, Tsien C, Dhermain F, Soffietti R, Mehta MP, Weller M, Tonn JC. Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients - a report of the PET/RANO group. Neuro Oncol. 2021 Jun 1;23(6):881-893. doi: 10.1093/neuonc/noab013. PMID 33538838
- [Background] Henderson F Jr, Brem S, O'Rourke DM, Nasrallah M, Buch VP, Young AJ, Doot RK, Pantel A, Desai A, Bagley SJ, Nabavizadeh SA. 18F-Fluciclovine PET to distinguish treatment-related effects from disease progression in recurrent glioblastoma: PET fusion with MRI guides neurosurgical sampling. Neurooncol Pract. 2020 Mar;7(2):152-157. doi: 10.1093/nop/npz068. Epub 2019 Dec 8. PMID 32206320
- [Background] Galldiks N, Langen KJ, Holy R, Pinkawa M, Stoffels G, Nolte KW, Kaiser HJ, Filss CP, Fink GR, Coenen HH, Eble MJ, Piroth MD. Assessment of treatment response in patients with glioblastoma using O-(2-18F-fluoroethyl)-L-tyrosine PET in comparison to MRI. J Nucl Med. 2012 Jul;53(7):1048-57. doi: 10.2967/jnumed.111.098590. Epub 2012 May 29. PMID 22645298
- [Background] Banerjee A, Jakacki RI, Onar-Thomas A, Wu S, Nicolaides T, Young Poussaint T, Fangusaro J, Phillips J, Perry A, Turner D, Prados M, Packer RJ, Qaddoumi I, Gururangan S, Pollack IF, Goldman S, Doyle LA, Stewart CF, Boyett JM, Kun LE, Fouladi M. A phase I trial of the MEK inhibitor selumetinib (AZD6244) in pediatric patients with recurrent or refractory low-grade glioma: a Pediatric Brain Tumor Consortium (PBTC) study. Neuro Oncol. 2017 Aug 1;19(8):1135-1144. doi: 10.1093/neuonc/now282. PMID 28339824
- [Background] Hutterer M, Nowosielski M, Putzer D, Jansen NL, Seiz M, Schocke M, McCoy M, Gobel G, la Fougere C, Virgolini IJ, Trinka E, Jacobs AH, Stockhammer G. [18F]-fluoro-ethyl-L-tyrosine PET: a valuable diagnostic tool in neuro-oncology, but not all that glitters is glioma. Neuro Oncol. 2013 Mar;15(3):341-51. doi: 10.1093/neuonc/nos300. Epub 2013 Jan 17. PMID 23335162
- [Background] Gelfand MJ. Dosimetry of FDG PET/CT and other molecular imaging applications in pediatric patients. Pediatr Radiol. 2009 Feb;39 Suppl 1:S46-56. doi: 10.1007/s00247-008-1023-6. Epub 2008 Dec 16. PMID 19083225
- [Background] Quinn BM, Gao Y, Mahmood U, Pandit-Taskar N, Behr G, Zanzonico P, Dauer LT. Patient-adapted organ absorbed dose and effective dose estimates in pediatric 18F-FDG positron emission tomography/computed tomography studies. BMC Med Imaging. 2020 Jan 29;20(1):9. doi: 10.1186/s12880-020-0415-4. PMID 31996149